CLINICAL TRIAL: NCT07343752
Title: Does Adding Blood Flow Restriction Training to the Physical Therapy Program Improve Outcomes in Adolescents With Spasmodic Flatfoot Deformity?
Brief Title: To Evaluate the Efficiency and Results of Adding BFR to the Physical Therapy Program fo Managing Adolescents Presented With Spasmotic Flatfoot Deformities Compared to the Standard Physical Therapy Program Without BFR
Acronym: BFR SFFD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam ibrahim, Physical tharapist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-2025-300682
Record Dates: First submitted 2025-12-02; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Flat Foot; Spastic
MeSH Terms: conditions — Flatfoot; Muscle Spasticity | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR (Experimental): Adding BFR to traditional low-intensity training.
  Interventions: Device: blood flow restriction
- control (No Intervention): traditional training

INTERVENTIONS:
Device: blood flow restriction — The addition of BFR to low-load dynamic exercise training is effective for augmenting changes in both muscle strength and size.
  Arms: BFR

SUMMARY:
The goal of this randomized clinical trial is to evaluate the efficiency and results of adding blood flow restriction (BFR) training to the physical therapy program for managing adolescents presented with spasmotic flatfoot deformities compared to the Standard physical therapy program without blood flow restriction.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents presented with idiopathic, rigid, spasmodic flatfeet.
* Age should be younger than 18 years old. 3- Patients who did not respond to initial medical treatment for three weeks.

Exclusion Criteria:

* generalised tarsal arthritis
* neurological disorder.
* secondary rigid flatfoot deformity
* patients who did not complete the follow up or evaluation protocol
* Patients who will refuse to participate

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle score (AOFAS) | baseline and 2 months
  Ankle-Hindfoot Scale: a standard method of reporting the clinical and functional status of the ankle and foot.
  The systems incorporate both subjective and objective factors into numerical scales to describe function, alignment, and pain. A score of 100 points is possible in a patient with no pain, full range of sagittal and hindfoot motion, no ankle or hindfoot instability, good alignment, ability to walk more than six blocks, ability to ambulate on any walking surface, no discernible limp, no limitation of daily or recreational activities, and no assistive devices needed for ambulation. Fifty points were assigned to function, 40 to pain, and 10 to alignment.
Range of motion (ROM) | baseline and at last follow up, 2 months
  Ankle range of motion of the sagittal plane (dorsiflexion and plantar flexion) and in the coronal plane (inversion and eversion), using a goniometer.

SECONDARY OUTCOMES:
Muscle power | baseline and at last follow up, 2 months
  Muscle power by dynamometer for: Tibialis anterior and Toe flexors
Numerical Pain Rating Scale (NPRS). | baseline and at last follow-up, 2 months
  Pain level using NPRS, a scale from 0 to 10, where 0 indicates no pain and 10 represents the worst pain imaginable.
Patient satisfaction | last follow up, 2 months
  Patient satisfaction: patient satisfaction was initially collected by a simple yes or no question and if they were willing to go through the same protocol again and if they were satisfied with the results followed by detailed measurements using the 0 to 10 scale reported by Park et al., where 0 is extremely unsatisfied, and 10 is extremely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Physical Therapy Unit, Asyut, Egypt